CLINICAL TRIAL: NCT04647656
Title: Hyperbaric Oxygen Therapy for Post-COVID-19 Syndrome: a Prospective, Randomized, Double Blind Study.
Brief Title: Hyperbaric Oxygen Therapy for Post-COVID-19 Syndrome
Acronym: HBOTpCOVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 332-20-ASF
Record Dates: First submitted 2020-11-29; First posted 2020-12-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Covid19; Neurocognitive Dysfunction
MeSH Terms: conditions — COVID-19; Cognition Disorders | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBOT treatment group (Active Comparator): 40 daily hyperbaric oxygen treatment sessions will be administered 5 days per week
  Interventions: Device: Hyperbaric oxygen
- HBOT sham group (Sham Comparator): 40 daily Sham non-hyperbaric oxygen treatment will be administered 5 days per week
  Interventions: Device: Sham

INTERVENTIONS:
Device: Hyperbaric oxygen — Each session will include exposure of 90 minutes to 100% at 2 ATA, with 5 minutes air breaks every 20 minutes
  Arms: HBOT treatment group
Device: Sham — Each session will include exposure of 90 minutes to 21% at 1.2 ATA during the first five minutes of the session with the noise of circulating air, and then decrease slowly during the next five minutes to 1.03 ATA
  Arms: HBOT sham group

SUMMARY:
Post-COVID-19 syndrome is an assembly of symptoms, following an infection with Coronavirus disease 2019 (COVID-19). The syndrome is characterized by cognitive impairment, fatigue, sleep disorders, smell and taste disorders, pain and more. This long-term sequela can last for months after recovering from the virus, and no treatment is known to date. The aim of this study is to compare the effect of HBOT vs. Sham on post COVID-19 syndrome

DETAILED DESCRIPTION:
Post-COVID-19 syndrome is an assembly of signs and symptoms first described on patients recovering from severe Coronavirus 2019 (COVID-19) infection. The syndrome is characterized by cognitive impairment, fatigue, and other neurologic symptoms. With time, and the growing understanding on this unique virus, there is cumulative case series reports on patients with mild to moderate disease, suffering from long standing post-COVID-19 syndrome. Taking in consideration, this pandemic is worldwide and still spreading, there's an urgent need for effective treatment for those patients who are suffering from the long standing, life debilitating, post-COVID-19 syndrome.

Neurologic signs and symptoms are common during hospitalization with COVID-19, with 42% of patients at onset of the disease and 82% during the course of the disease. Patients report mainly on myalgias, headaches, encephalopathy, dizziness, dysgeusia, and anosmia. After recovering from COVID-19, many patients continue to suffer from symptoms. Only 13% of the patients were completely free of symptoms after full resolution of the virus. The main symptom, reported by more than half the patients included cognitive impairment, fatigue and sleep disorders. A recent study analyzed data from 84,285 Individuals who recovered from suspected or confirmed COVID-19 showed reduced cognitive performance. This deficit scales with symptom severity and is evident amongst those without hospital treatment.

Two main biological sequelae of COVID-19 might play a role in the pathogenesis of this syndrome. The first is hypercoagulability state accompanies acute infection. This is characterized by increased risk of small and large vessel occlusion and is associated with increased mortality [9]. Neurologic complications might be a result of micro-infarcts in the central of peripheral nervous system; The second is an uncontrolled inflammatory response, called cytokines storm. This cytokine release is characterized by an increase in interleukin (IL)-1, IL-6, tumor necrosis factor (TNF)-α and a change in macrophages population. Thus, COVID-19 can cause neuroinflammation, that might be prolonged and lead to signs of post-COVID-19 syndrome.

The Micro-infarcts and neuroinflammation are important causes of local hypoxia, and specifically neurological hypoxia. One of the options to reverse hypoxia, reduce neuroinflammation and induce neuroplasticity is hyperbaric oxygen therapy (HBOT).

Hyperbaric oxygen therapy (HBOT) includes the inhalation of 100% oxygen at pressures exceeding 1 atmosphere absolute, thus enhancing the amount of oxygen dissolved in the body tissues. During HBOT, the arterial O2 tension typically exceeds 2000 mmHg, and levels of 200-400 mmHg occur in tissues Even though many of the beneficial effects of HBOT can be explained by improvement of tissue oxygenation, it is now understood that the combined action of hyperoxia and hyperbaric pressure, triggers both oxygen and pressure sensitive genes, resulting in inducing regenerative processes including stem cells proliferation and mobilization with anti-apoptotic and anti-inflammatory factors.

The HBOT protocol will be administrated in a multi-place chamber. The protocol includes 40 daily sessions, 5 sessions per week for two months. Treatment group will subjected to 100% oxygen by mask at 2 atmosphere (ATA) for 90 minutes with 5 minute air breaks every 20 minutes. Sham group will be subjected to 21% oxygen by mast for 90 minutes, at 1.2 ATA during the first five minutes of the session with the noise of circulating air, and then decrease slowly during the next five minutes to 1.03 ATA.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Reported post COVID-19 cognitive deterioration that effect quality of life and persist at least 3 months after confirmed infection.
3. Subject willing and able to read, understand and sign an informed consent

Exclusion Criteria:

1. Inability to attend scheduled clinic visits and/or comply with the study protocol
2. History of traumatic brain injury (TBI) or any other non COVID brain pathology
3. Active malignancy
4. Substance use at baseline
5. Severe or unstable physical disorders or major cognitive deficits at baseline
6. HBOT for any reason prior to study enrolment
7. Chest pathology incompatible with pressure changes (including moderate to severe asthma)
8. Ear or Sinus pathology incompatible with pressure changes
9. An inability to perform an awake brain MRI
10. Active smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Cognitive health assessment (NeuroTrax) | Baseline, 2 months
  Memory, attention and information process will be evaluated using the NeuroTrax computerized cognitive evaluation battery.

SECONDARY OUTCOMES:
Brain perfusion | Baseline, 2 months
  Cerebral blood volume and flow will be measured using perfusion MRI protocol Dynamic susceptibility contrast (DSC).
Brain microstructure Brain microstructure | Baseline, 2 months
  Fractional anisotropy (FA) and Mean diffusivity (MD) will be evaluated using diffusion tensor imaging (DTI) MRI protocol
Brain function imaging | Baseline, 2 months
  Resting state fMRI (rsfMRI), and task based fmri will evaluate brain function during a working memory task
Post-COVID-19 symptom | Baseline, 2 months
  Self-reported questionnaire covers the most common symptoms related to post-coronavirus 2019 (COVID-19) disease
Quality of Life SF-36 | Baseline, 2 months, 1 year
  Short Form (SF)-36 questionnaire for self reporting quality of life
The Pittsburgh Sleep Quality Index PSQI | Baseline, 2 months, 1 year
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality
The Brief Symptom Inventory - 18 (BSI-18) | Baseline, 2 months, 1 year
  The BSI-18 will be used to evaluate psychological distress. The BSI-18 is an 18 item self-report questionnaire which generates a summary scale, the global stress index (GSI), and three subscales: depression, anxiety, and somatization
BPI - Brief pain inventory (short form) | Baseline, 2 months, 1 year
  The Brief pain inventory (BPI) is a short, self-administered questionnaire. It contains 15 items, which include 2 multi-item scales measuring pain intensity and the impact of pain on functioning and well-being.
Neuro-physical evaluation | Baseline, 2 months
  Static balance will be assessed by the Balance Error Scoring System (BESS); Dynamic balance and risk of falling will be assessed by the Timed Up and Go test (TUG) and 10-meter walk (10MW).
  Muscle function will be assessed by the sit to stand (STS) test for the leg strength and endurance and hand-held dynamometry (HHD) for the isometric grip strength.
  The sub-maximal aerobic capacity and endurance will be assessed by the 6-minute walk test (6MWT).
Neurological evaluation | Baseline, 2 months
  The neurological exam will include tests of the cranial nerves, motor, sensory and cerebellar function and gait
Smell and taste evaluations. | Baseline, 2 months
  Smell will be tested through smell identification kits to test for odour detection, discrimination and threshold. The kit is standardized for age and gender, and available in different languages (Sniffing sticks).
  Taste will be tested on bilateral anterior and posterior parts of the tongue by four tastes: bitter, sour, salt and sweet ("The Taste Strip Test").
Cardiopulmonary exercise test | Baseline, 2 months
  The cardiopulmonary exercise test (CPET) is a non-invasive measurement of the cardiovascular system, respiratory system and muscles.
Echocardiography | Baseline, 2 months
  Conventional echocardiography evaluation, linear, volumetric and Doppler measurements will be performed to assess cardiac functions.
Lung functions test | Baseline, 2 months
  Measurements of pulmonary functions will be performed using spirometry (the MiniSpir) testing apparatus.
Immune system | Baseline, 2 months
  Blood tests will evaluate immune system including cytokines, c-reactive protein (CRP) and COVID-19 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Shai a Efrati, MD, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Assaf-Harofeh medical center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stam HJ, Stucki G, Bickenbach J; European Academy of Rehabilitation Medicine. Covid-19 and Post Intensive Care Syndrome: A Call for Action. J Rehabil Med. 2020 Apr 15;52(4):jrm00044. doi: 10.2340/16501977-2677. PMID 32286675
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Garrigues E, Janvier P, Kherabi Y, Le Bot A, Hamon A, Gouze H, Doucet L, Berkani S, Oliosi E, Mallart E, Corre F, Zarrouk V, Moyer JD, Galy A, Honsel V, Fantin B, Nguyen Y. Post-discharge persistent symptoms and health-related quality of life after hospitalization for COVID-19. J Infect. 2020 Dec;81(6):e4-e6. doi: 10.1016/j.jinf.2020.08.029. Epub 2020 Aug 25. PMID 32853602
- [Background] Tal S, Hadanny A, Berkovitz N, Sasson E, Ben-Jacob E, Efrati S. Hyperbaric oxygen may induce angiogenesis in patients suffering from prolonged post-concussion syndrome due to traumatic brain injury. Restor Neurol Neurosci. 2015;33(6):943-51. doi: 10.3233/RNN-150585. PMID 26484702
- [Background] Boussi-Gross R, Golan H, Fishlev G, Bechor Y, Volkov O, Bergan J, Friedman M, Hoofien D, Shlamkovitch N, Ben-Jacob E, Efrati S. Hyperbaric oxygen therapy can improve post concussion syndrome years after mild traumatic brain injury - randomized prospective trial. PLoS One. 2013 Nov 15;8(11):e79995. doi: 10.1371/journal.pone.0079995. eCollection 2013. PMID 24260334
- [Derived] Leitman M, Fuchs S, Tyomkin V, Hadanny A, Zilberman-Itskovich S, Efrati S. The effect of hyperbaric oxygen therapy on myocardial function in post-COVID-19 syndrome patients: a randomized controlled trial. Sci Rep. 2023 Jun 10;13(1):9473. doi: 10.1038/s41598-023-36570-x. PMID 37301934